CLINICAL TRIAL: NCT02237066
Title: Understanding the Mechanism of Peripheral Arterial Balloon Angioplasty by the Chocolate PTA Balloon Catheter Compared to Conventional PTA Balloons Via OCT Imaging
Brief Title: Understanding Angioplasty by the Chocolate PTA Balloon Catheter Compared to Conventional PTA Balloons Via OCT Imaging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment goals were not able to be met
Sponsor: TriReme Medical, LLC (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chocolate OCT
Record Dates: First submitted 2014-09-03; First posted 2014-09-11 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Infrainguinal Peripheral Arterial Disease
Keywords: OCT; PTA; Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chocolate PTA Balloon (Experimental): Chocolate PTA Balloon Angioplasty
  Interventions: Device: Chocolate PTA Balloon Angioplasty
- Standard PTA Balloon (Active Comparator): Standard PTA Balloon Angioplasty
  Interventions: Device: Standard PTA Balloon Angioplasty

INTERVENTIONS:
Device: Chocolate PTA Balloon Angioplasty — OCT imaging of diseased vessel is treated with an Angioplasty Procedure using the Chocolate PTA Balloon Catheter followed by OCT imaging of the treated area immediately after balloon use and 10 minutes later
  Arms: Chocolate PTA Balloon
Device: Standard PTA Balloon Angioplasty — OCT imaging of diseased vessel is treated with an Angioplasty Procedure using a standard PTA Balloon Catheter followed by OCT imaging of the treated area immediately after balloon use and 10 minutes later
  Arms: Standard PTA Balloon

SUMMARY:
The purpose of this study is to compare the Chocolate PTA Balloon to standard Percutaneous Transluminal Angioplasty (PTA) catheters. The investigators will use Optical Coherence Tomography (OCT) and Quantitative Vascular Angiography to evaluate the acute vascular response of vessels treated with the Chocolate Balloon to a standard balloon catheter, with the primary endpoint being luminal gain assessed by OCT lumen volume measurements.

DETAILED DESCRIPTION:
Subjects will be randomized to treatment with either the Chocolate Balloon catheter or a standard balloon angioplasty catheter. All angioplasty procedures will be conducted with treatment balloon at the full discretion of the physician and according to the standard practice at the hospital and the device Instructions for Use. All patients will undergo baseline OCT imaging in addition to standard angiography. Post-PTA, all patients will then undergo repeat OCT imaging immediately post-procedure and then again at 10-minutes post-procedure to assess for vascular recoil.

ELIGIBILITY:
Inclusion Criteria:

* Reference Vessel Diameter (RVD) between 2.5 and 6.0mm and within treatment range of available balloon at Target Lesion
* Intermittent claudication or critical limb ischemia (Rutherford 3-5)
* De novo stenosis (≥70%) or occlusion in the infrainguinal arteries, including superficial femoral artery (SFA), popliteal, and infrapopliteal arteries.
* Lesion successfully crossed with a guide-wire
* Patient has given informed consent to participate in this study

Exclusion Criteria:

* Lesion requiring ablative procedures (i.e. atherectomy or laser) as part of treatment
* Lesion length >75mm
* Previous bypass or stent at target vessel or proximal to target vessel
* Significant in-flow disease at target lesion
* Known inadequate distal outflow disease or planned treatment of vessel distal to target lesion
* Acute limb ischemia or need for thrombolytic therapy
* Known intolerance to required study medications, contrast media, or nitinol
* Known impaired Renal Function with Glomerular Filtration Rate (GFR) <45 ml/min per 1.73m2
* Known bleeding disorder or uncontrolled hypercoagulable disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Luminal Gain | Average of 90 minutes
  Luminal Gain as defined by OCT lumen volume measurements. Luminal gain is assessed as the percentage change comparing pre-treatment and post-treatment volume measurements in cubic centimeters (CC) or millimeters (m3).

SECONDARY OUTCOMES:
Dissection | Average of 90 minutes
  Dissection severity (extension) as defined by both angiographic and OCT metrics.
  Dissections occur when the blood goes into the vessel wall instead of staying in the vessel lumen. Dissection severity is determined by a visual review of the angiogram and OCT images by an independent core lab. Dissections are classified as flow-limiting (more severe) vs. non-flow limiting (less severe) based upon the amount of the blood that is flowing into the vessel wall.
Hematoma | Average of 90 minutes
  Presence of intramural hematoma on OCT.
  A hematoma can be visually observed on a angiogram and an OCT image. The images will be independently reviewed by a core lab expert who will document if a hematoma is present or not.
Optimal PTA | Average of 90 minutes
  Achievement of Optimal PTA (<30% Diameter stenosis without flow limiting dissection)
  <30% Diameter stenosis and flow limiting dissections are visual assessments that will be conducted by an independent core lab review. The % diameter stenosis measures the amount of plaque that is in the vessel and a flow-limiting dissection is observed as either present or not present.

CONTACTS AND LOCATIONS:
Overall Officials: Sahil A Parikh, MD, Principal Investigator — Harrington Heart and Vascular Institute University Hospitals Case Medical Center
Locations (2):
- United States (2):
  - Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio